CLINICAL TRIAL: NCT02420977
Title: Evaluation of PSMA-based PET as an Imaging Biomarker of Androgen Receptor Signaling in High-Risk Localized and Locally Advanced Prostate Cancer
Brief Title: Evaluation of PSMA-based PET as an Imaging Biomarker in Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1560; IRB00065395 (Other: JHM IRB); 1U01CA183031-01A1 (NIH)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Advanced Prostate Cancer
Keywords: radiotracer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DCFPyL PET-MRI fusion or PET/MRI (Experimental): * Pelvic DCFPyL PET-MRI fusion or PET/MRI compared before and after 2-3 months of ADT
  * Pelvic DCFPyL PET-MRI fusion or PET/MRI compared before and after 2-3 months
  Interventions: Drug: Pelvic DCFPyL PET-MRI fusion or PET/MRI

INTERVENTIONS:
Drug: Pelvic DCFPyL PET-MRI fusion or PET/MRI — * Pelvic DCFPyL PET-MRI fusion or PET/MRI compared before and after 2-3 months of ADT
  * Pelvic DCFPyL PET-MRI fusion or PET/MRI compared before and after 2-3 months

SUMMARY:
This research is being done to see if an investigational radioactive imaging agent (radiotracer) called 18F-DCFPyL can help us find prostate cancer at its original site in the prostate gland and in distant sites (bone, lymph nodes) in men diagnosed with prostate cancer before surgery.

DETAILED DESCRIPTION:
The investigators propose to evaluate the feasibility of using a novel small molecule PET radiotracer, DCFPyL to target prostate cancer prostate-specific membrane antigen (PSMA). PSMA is a well studied cell surface marker of prostate cancer with increased expression associated with higher tumor grade and advanced metastatic tumors. More specifically it is associated with a higher Gleason score and there is evidence it can serve as a potential marker for prostate tumor carcinogenesis, progression and as a AR signaling surrogate marker of ADT response. This small molecule PET radiotracer specifically targeting an important prostate specific marker of AR signaling dynamics following ADT, tumor progression and metastatic potential warrants validation as an in-vivo non-invasive imaging biomarker for PSMA expression and prostate cancer detection.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years of age or greater with recently diagnosed prostate cancer with planned radiation and ADT.
* Key inclusion criteria (the entire list of inclusion and exclusion criteria will appear later in section 4 of the protocol)

  * Newly diagnosed prostate cancer pathologically proven by prostate biopsy
  * Prostate biopsy histology grade ≥ Gleason 8-10
  * Patients considered as candidates for and medically fit to undergo radiation and ADT
  * At least 10 days after most recent prostate biopsy

Exclusion Criteria:

* Prior pelvic external beam radiation therapy or brachytherapy
* Chemotherapy for prostate cancer
* Hormone deprivation therapy
* Investigational therapy for prostate cancer
* Hemorrhagic cystitis or active prostatitis

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Response rate differences | baseline and after 2-3 months
  To compare the detection , sextant localization and response of DCFPyL PET-MRI fusion or PET/MRI before and after 2-3 months of ADT in men with biopsy-positive high-risk localized or locally advanced prostate cancer.

SECONDARY OUTCOMES:
Biomarker changes | Baseline and at 2=3 months
  To compare DCFPyL PET-MRI fusion or PET/MRI uptake in prostate cancer (quantified as per sextant SUVmax, SUVavg, metabolic tumor volume, total lesion DCFPyL uptake, DCFPyL uptake rate) as a reliable non-invasive imaging biomarker of PSMA expression following ADT as determined by qualitative and quantitative MRI-guided prostate biopsy core tissue immunohistochemical analysis. DCFPyL uptake will also be compared to other prostate cancer relevant marker expression levels (PSA, Ki-67, TMPRSS2-ERG) by immunohistochemical analysis.
Metabolic tumor uptake changes | baseline and then at 2-3 months
  To compare DCFPyL PET-MRI fusion or PET/MRI uptake in primary prostate cancer (quantified as per sextant SUVmax, SUVavg, metabolic tumor volume, total lesion DCFPyL uptake, DCFPyL uptake rate) following ADT with standard clinical prognostic markers (PSA, Gleason score, clinical stage) and with predictive model of pathologic stage.
Gene expression changes | Baseline and then at 2-3 months
  To validate DCFPyL PET-MRI fusion or PET/MRI uptake in prostate cancer (quantified as per sextant SUVmax, SUVavg, metabolic tumor volume, total lesion DCFPyL uptake, DCFPyL uptake rate) as a reliable non-invasive imaging biomarker of AR signaling following ADT as determined by AR gene set expression of biopsy core tissue specimens using qPCR.
Nodal metastatic disease changes | Baseline and then at 2-3 months
  To compare the detection of nodal metastatic disease by DCFPyL PET-MRI fusion or PET/MRI at initial staging to detection by available conventional imaging modalities (bone scan, CT, MRI) and when available biopsy pathology.
All cause DCFPyL PET-MRI fusion or PET/MRI toxicity | Baseline and then at 2-3 months
  To determine the safety of DCFPyL.

CONTACTS AND LOCATIONS:
Overall Officials: Curtiland Deville, M.D., Principal Investigator — The SKCCC at Johns Hopkins
Locations (1):
- Curtiland Deville, Baltimore, Maryland, United States